CLINICAL TRIAL: NCT03229759
Title: A Randomized Single Center Blinded Clinical Evaluation of the Antimicrobial Effectiveness of an Antimicrobial Cloth Compared to Vehicle and 0.9% Saline
Brief Title: Evaluation of the Antimicrobial Effectiveness of an Antimicrobial Cloth
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MPS-17IPVAW10
Record Dates: First submitted 2017-07-17; First posted 2017-07-26 (Actual); Results first posted 2021-04-23 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-03

CONDITIONS: Preoperative Skin Preparation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Investigational Product (Experimental): Polyester cloth impregnated with investigational product
  Interventions: Drug: Octenidine Dihydrocloride in aqueous solution
- Vehicle Control (VC) (Placebo Comparator): Polyester cloth impregnated with the vehicle control
  Interventions: Other: Vehicle Control
- Saline Control (SC) (Placebo Comparator): Saline applied wtih polyester cloth
  Interventions: Other: Saline Control

INTERVENTIONS:
Drug: Octenidine Dihydrocloride in aqueous solution — application of investigational product
  Arms: Investigational Product
Other: Vehicle Control — application of vehicle control
  Arms: Vehicle Control (VC)
Other: Saline Control — application of placebo
  Arms: Saline Control (SC)

SUMMARY:
Healthy volunteers will receive treatment to two body locations with the investigational product and placebo and the antimicrobial effectiveness of each treatment will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Males and/or females, at least 18 years or older and of any race.
* Are in good general health.
* Unable to become pregnant, or willing to use an acceptable method of contraception (i.e. oral contraception, intra-uterine device [IUD], diaphragm, condom, abstinence, bilateral Tubal ligation, or are in a monogamous relationship with a partner who has had a Vasectomy) to prevent pregnancy for at least 14 days immediately preceding Treatment Day and throughout the duration of the study, if female of child-bearing potential.
* All female subjects must have a negative urine pregnancy test on Treatment Day prior to any applications of the study products.
* Have skin within 6 inches of the test sites that is free of dermatoses, abrasions, cuts, lesions or other skin disorders.
* Cooperative and willing to follow Subject Instructions
* Cooperative and willing to sign Consent Form and HIPAA Authorization Form.
* Able to read, write and follow instructions in English.

Exclusion Criteria:

* Exposure to topical or systemic antimicrobials or any other product known to affect the normal microbial flora of the skin, antibiotics or steroids (other than hormones for contraception or post-menopausal reasons) exposure within 14 days prior to Treatment Day and for the remainder of the study. Restrictions include, but are not limited to antimicrobial-containing soaps, antiperspirants/deodorants, shampoos, lotions, perfumes, after shaves, and colognes.
* Swimming in chemically treated pools or bathing in hot tubs, spas and whirlpools within 14 days prior to Treatment Day and for the remainder of the study.
* Use of tanning beds, hot waxes, or depilatories, including shaving (in the applicable test areas) within 14 days prior to Treatment Day and for the remainder of the study.
* Contact with strong detergents, solvents, acids, bases, bug repellant, fabric softener-treated clothing, UV treated clothing or other household chemicals in the applicable test areas within 14 days of the Treatment Day and for the remainder of the study.
* Subjects who have a history of sensitivity to vinyl, natural rubber latex, adhesive skin products (e.g., Band-Aids, medical tapes), polyester, metals, inks, common antibacterial agents found in common personal beauty or personal care soaps, lotions, or ointments
* Subjects who have asthma requiring medication, diabetes, hepatitis B or C, an organ transplant, mitral valve prolapse with a heart murmur, congenital heart disease, lupus, Crohn's disease, medicated multiple sclerosis, internal prosthesis or any immunocompromised conditions (such as AIDS or HIV positive).
* Subjects who have a history of skin allergies.
* Subjects who have a history of skin cancer within 6 inches of the applicable test areas or have received treatment for any type of internal cancer within the 5 years prior to enrollment.
* Any tattoos or scars on the test sites or within 2 inches of the test sites; skin blemishes or warts may be permissible with the specific approval of the Principal Investigator or consulting physician.
* Dermatoses, cuts, lesions, active skin rashes, scabs, breaks in the skin or other skin disorders within 6 inches on or around the test sites.
* A currently active skin disease or inflammatory skin condition (for example contact dermatitis; psoriasis, and eczema) anywhere on the body.
* Subjects who are pregnant, attempting pregnancy, or nursing.
* Subjects who have showered or bathed within at least 72 hours of the Treatment Day (sponge baths may be taken, however, the lower abdomen and upper thigh region must be avoided).
* Subjects who receive an irritation score of 1 (any redness, swelling, rash, or dryness present at any treatment area) for any individual skin condition prior to the Treatment Day baseline sample collection.
* Participation in another clinical trial in the 30 days prior to signing the informed consent for this study, current enrollment in another clinical trial, or have already participated in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2017-08-04 (Actual); Study Completion 2017-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Beausoleil, Principal Investigator — BioScience Laboratories
Locations (1):
- BioScience Laboratories, Bozeman, Montana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were only treated if baseline bacterial counts met the inclusion criteria.
  Participants were treated with 2 of 3 study products (Investigational Product, saline control, vehicle control) 1 on the left side of the body (both groin and abdomen), 1 on the right side of the body (both groin and abdomen). Therefore, treatment groups are not discrete categories.
Groups:
- All Participants: All screened participants
Period: Overall Study
Arm/Group | All Participants
Started (Participants consented and enrolled.) | 99
Participants Treated | 69
Treated With Investigational Product (Participants were treated with 2 of 3 study products.) | 45
Treated With Vehicle Control (Participants were treated with 2 of 3 study products.) | 47
Treated With Saline Control (Participants were treated with 2 of 3 study products.) | 46
Completed | 69
Not Completed | 30
Not completed — Screen Failure | 30

BASELINE CHARACTERISTICS:
Population: Participants were treated with multiple study products. Therefore, treatment groups are not discrete categories and cannot be displayed by treatment group.
Groups:
- Participants Treated: Participants who received study product at at least 1 treatment site (abdomen and/or groin). Participants were treated with 2 of 3 study products, investigational product (IP), saline control (SC), and/or vehicle control (VC). Therefore, treatments arms are not discrete groups of participants. Therefore, baseline data are presented for all treated participants and not by treatment arm.
Arm/Group | Participants Treated
Number analyzed (Participants) | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 63
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 64
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 69

OUTCOME MEASURES:

1. Primary Outcome: Bacterial Count at 10 Minutes Post Application
Time Frame: 10 minutes after application of test product
Population: Analysis only includes participants with required treatment day baseline bacterial counts at each anatomical site at baseline and non-missing data at 10 minutes.
Measure: Mean (Standard Deviation); unit: log10 CFU/cm^2
Groups:
- Investigational Product: Investigational Product (IP) - Thermally treated polyester cloths impregnated with 0.4% weight by volume octenidine dihydrochloride (OCT) aqueous solution
- Saline Control: Saline Control (SC) - 0.9% saline applied with polyester cloths
- Vehicle Control: Vehicle Control (VC) Thermally treated polyester cloths impregnated with vehicle formulation.
Arm/Group | Investigational Product | Saline Control | Vehicle Control
Number analyzed (Participants) | 41 | 41 | 42
log10 CFU/cm^2
  Abdomen- Baseline: number analyzed (Participants) | 28 | 29 | 26
  Abdomen- Baseline | 3.55 (0.40) | 3.61 (0.41) | 3.66 (0.40)
  Abdomen- 10 minutes: number analyzed (Participants) | 28 | 29 | 26
  Abdomen- 10 minutes | 1.19 (1.28) | 2.64 (0.58) | 2.56 (0.97)
  Groin- Baseline: number analyzed (Participants) | 31 | 26 | 28
  Groin- Baseline | 5.95 (0.60) | 6.07 (0.53) | 5.89 (0.47)
  Groin- 10 minutes: number analyzed (Participants) | 31 | 26 | 28
  Groin- 10 minutes | 2.98 (1.14) | 4.90 (0.56) | 4.25 (0.68)
Statistical Analysis 1: Comparison: Investigational Product vs Saline Control; Test on abdomen Average treatment effect was calculated using a linear regression model for each body site was used for primary analysis. In the model, the response was the post-treatment log10 bacterial counts and predictors were the treatment effect as a fixed effect and the pre-treatment log10 bacterial counts as a covariate; Test type: Superiority; Mean Difference (Final Values) = 1.48, 95% CI 2-sided [0.88 to 2.08]
Statistical Analysis 2: Comparison: Investigational Product vs Vehicle Control; Tested on the abdomen Analysis was performed based on deferral letters from the FDA. Average treatment effect was calculated using a linear regression model for each body site was used for primary analysis. In the model, the response was the post-treatment log10 bacterial counts and predictors were the treatment effect as a fixed effect and the pre-treatment log10 bacterial counts as a covariate; Test type: Superiority; Mean Difference (Final Values) = 1.34, 95% CI 2-sided [0.72 to 1.96]
Statistical Analysis 3: Comparison: Investigational Product vs Saline Control; Groin; Test type: Superiority; Mean Difference (Final Values) = 1.93, 95% CI 2-sided [1.38 to 2.47]
Statistical Analysis 4: Comparison: Investigational Product vs Vehicle Control; Groin; Test type: Superiority; Mean Difference (Final Values) = 1.26, 95% CI 2-sided [0.73 to 1.79]

ADVERSE EVENTS:
Time Frame: 10 minutes
Groups:
- Subject Treated: Participants who received study product at at least 1 treatment site (abdomen and/or groin). Participants were treated with 2 of 3 study products, investigational product (IP), saline control (SC), and/or vehicle control (VC). Therefore, treatments arms are not discrete groups of participants. Therefore, adverse event data are presented for all treated participants and not by treatment arm.
Arm/Group | Subject Treated
All-Cause Mortality (participants affected / at risk) | 0/69
Serious Adverse Events (participants affected / at risk) | 0/69
Other Adverse Events (participants affected / at risk) | 0/69

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-05-25): https://cdn.clinicaltrials.gov/large-docs/59/NCT03229759/Prot_001.pdf
  • Statistical Analysis Plan (2017-06-23): https://cdn.clinicaltrials.gov/large-docs/59/NCT03229759/SAP_002.pdf